CLINICAL TRIAL: NCT03438682
Title: Real World Effectiveness and Safety of Hysteroscopic (Essure®) Compared to Laparoscopic Sterilization
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: University of California, Davis (Other); National Center for Health Research (Unknown); Patient-Centered Outcomes Research Institute (Other); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2000020734; 1U01FD005938-01 (FDA)
Record Dates: First submitted 2018-01-29; First posted 2018-02-20 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Sterility, Female; Contraception; Contraceptive Device; Complications
MeSH Terms: conditions — Infertility, Female | interventions — Intrauterine Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Essure Hysteroscopic Sterilization: Women who have undergone Essure hysteroscopic sterilization
  Interventions: Device: Essure
- Laparoscopic Sterilization: Women who have undergone laparoscopic sterilization
  Interventions: Procedure: Laparoscopic sterilization
- Intrauterine device (IUD) placement: Women who have undergone IUD placement
  Interventions: Device: Intrauterine Device (IUD)

INTERVENTIONS:
Device: Essure — Essure hysteroscopic sterilization
  Groups: Essure Hysteroscopic Sterilization
Procedure: Laparoscopic sterilization — Laparoscopic sterilization via electrocautery, ring, or clip.
  Groups: Laparoscopic Sterilization
Device: Intrauterine Device (IUD) — Intrauterine Device (IUD)
  Groups: Intrauterine device (IUD) placement

SUMMARY:
More than 345,000 U.S. women undergo either tubal ligation ("getting her tubes tied") or Essure procedures each year to permanently avoid pregnancy. Both prevent pregnancy by blocking women's Fallopian tubes but neither are 100% effective. Both can have complications, but not enough is known to help women make an informed choice between the two.

Essure is popular because it can be performed without anesthesia in a doctor's office and women can return to work the next day. However, patients have reported that the Essure procedure was unexpectedly painful. Also, women need to use other contraceptives for 3 months and then return for testing, to make sure their tubes are blocked and will prevent pregnancy. Not all women return for this test and some may get pregnant before realizing their Essure didn't work.

Essure was approved by the Food and Drug Administration (FDA) in 2002, but no studies ever compared it to tubal ligation. By 2015, over 9,000 women reported serious complications to the FDA. Women who were unhappy with Essure found each other online and created a Facebook "Essure Problems" support group that now has over 31,000 members. After an FDA Advisory Board expressed concerns about Essure's risks, in 2016 the FDA required stronger warnings about complications and announced that "more rigorous research" was needed, demanding Essure's maker conduct a new study comparing the benefits and risks of Essure to tubal ligation. Unfortunately, that study will not be finished before September 2023.

To provide answers as rapidly as possible for women considering sterilization, we will analyze data from the medical records of thousands of women with sterilization procedures funded by California's Medicaid. As poor women and women of color have different experiences with healthcare, and they more often choose sterilization, comparing these women's experiences with Essure and tubal ligation is very important. We will compare the safety and effectiveness of the 2 sterilization procedures to answer:

* How many women got pregnant afterwards?
* How many operations did each woman need to become infertile?
* Which complications did women have (i.e. chronic pain, depression)? We will also check whether certain women (such as certain age groups or those with diabetes) were most likely to have problems after either procedure.

DETAILED DESCRIPTION:
Study Aims:

Aim 1. To compare the real world effectiveness of hysteroscopic sterilization, laparoscopic sterilization and intrauterine devices (IUDs) by calculating:

1. Pregnancy rates at 3, 6, 12, 24, 36, 48, and 60 months post-procedure, indicating sterilization failure.
2. Patient's ability to rely on sterilization after hysteroscopic sterilization (blocked tubes on hysterosalpingogram) compared to laparoscopic sterilization and IUDs at 3, 6, 12, 24, 36, 48, and 60 months post-procedure, indicating concern of sterilization failure.

Aim 2. To compare safety and complications after hysteroscopic sterilization laparoscopic sterilization, and IUD placement by:

1. Evaluating rates of reoperation to achieve sterilization or reinsertion to achieve IUD placement at 3, 6, 12, 24, 36, 48, and 60 months post-procedure.
2. Evaluating other outcomes suggested by patient partners, including additional surgeries due to complications, chronic pain, and/or depression, by measuring claims for narcotic prescriptions, and antidepressants at 3, 6, 12, 24, 36, 48, 60 months post-procedure (hysteroscopic sterilization, laparoscopic sterilization, or IUD placement).
3. Identify sociodemographic and pre-sterilization clinical variables which may predict complications following hysteroscopic sterilization compared to laparoscopic sterilization and to IUDs.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-50 years at the time of sterilization procedure
* Claims indicating hysteroscopic or laparoscopic sterilization procedures or IUD placement

Exclusion Criteria:

* Active cancer
* Any conditions that would have excluded the patient for hysteroscopic sterilization
* Any conditions that would have excluded the patient for laparoscopic sterilization

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will use linked data from Centers for Medicare and Medicaid Services (CMS) Research Data Assistance Center (ResDAC) including research identifiable files (RIF) containing Medicaid records, known as the Medicaid Analytic Extract (MAX) files to identify women who have undergone hysteroscopic or laparoscopic sterilization procedures or IUD placement. The MAX files contain claims, encounters, and eligibility information on recipients of California's Medicaid program (Medi-Cal).
Sampling Method: Non-Probability Sample
Enrollment: 89203 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of hysteroscopic compared to laparoscopic sterilization and IUD placement (Aim 1a) | Pregnancy rates at 3 months post-procedure
  Pregnancy after sterilization or IUD placement, indicating failure
Effectiveness of hysteroscopic compared to laparoscopic sterilization and IUD placement (Aim 1a) | Pregnancy rates at 6 months post-procedure
  Pregnancy after sterilization or IUD placement, indicating failure
Effectiveness of hysteroscopic compared to laparoscopic sterilization and IUD placement (Aim 1a) | Pregnancy rates at 12 months post-procedure
  Pregnancy after sterilization or IUD placement, indicating failure
Effectiveness of hysteroscopic compared to laparoscopic sterilization and IUD placement (Aim 1a) | Pregnancy rates at 24 months post-procedure
  Pregnancy after sterilization or IUD placement, indicating failure
Effectiveness of hysteroscopic compared to laparoscopic sterilization and IUD placement (Aim 1a) | Pregnancy rates at 36 months post-procedure
  Pregnancy after sterilization or IUD placement, indicating failure
Effectiveness of hysteroscopic compared to laparoscopic sterilization and IUD placement (Aim 1a) | Pregnancy rates at 48 months post-procedure
  Pregnancy after sterilization or IUD placement, indicating failure
Effectiveness of hysteroscopic compared to laparoscopic sterilization and IUD placement (Aim 1a) | Pregnancy rates at 60 months post-procedure
  Pregnancy after sterilization or IUD placement, indicating failure

SECONDARY OUTCOMES:
Blocked fallopian tubes on post-procedure hysterosalpingogram test (Aim 1b) | 3 months post-procedure
  Ability to rely on sterilization after hysteroscopic sterilization (assessed by having blocked tubes on post-procedure hysterosalpingogram test) compared to laparoscopic sterilization and IUDs
Blocked fallopian tubes on post-procedure hysterosalpingogram test (Aim 1b) | 6 months post-procedure
  Ability to rely on sterilization after hysteroscopic sterilization (assessed by having blocked tubes on post-procedure hysterosalpingogram test) compared to laparoscopic sterilization and IUDs
Blocked fallopian tubes on post-procedure hysterosalpingogram test (Aim 1b) | 12 months post-procedure
  Ability to rely on sterilization after hysteroscopic sterilization (assessed by having blocked tubes on post-procedure hysterosalpingogram test) compared to laparoscopic sterilization and IUDs
Blocked fallopian tubes on post-procedure hysterosalpingogram test (Aim 1b) | 24 months post-procedure
  Ability to rely on sterilization after hysteroscopic sterilization (assessed by having blocked tubes on post-procedure hysterosalpingogram test) compared to laparoscopic sterilization and IUDs
Blocked fallopian tubes on post-procedure hysterosalpingogram test (Aim 1b) | 36 months post-procedure
  Ability to rely on sterilization after hysteroscopic sterilization (assessed by having blocked tubes on post-procedure hysterosalpingogram test) compared to laparoscopic sterilization and IUDs
Blocked fallopian tubes on post-procedure hysterosalpingogram test (Aim 1b) | 48 months post-procedure
  Ability to rely on sterilization after hysteroscopic sterilization (assessed by having blocked tubes on post-procedure hysterosalpingogram test) compared to laparoscopic sterilization and IUDs
Blocked fallopian tubes on post-procedure hysterosalpingogram test (Aim 1b) | 60 months post-procedure
  Ability to rely on sterilization after hysteroscopic sterilization (assessed by having blocked tubes on post-procedure hysterosalpingogram test) compared to laparoscopic sterilization and IUDs
Reoperation to achieve sterilization or reinsertion to achieve IUD placement | 3 months post-procedure
  Evaluating rates of reoperation to achieve sterilization or reinsertion to achieve IUD placement
Reoperation to achieve sterilization or reinsertion to achieve IUD placement | 6 months post-procedure
  Evaluating rates of reoperation to achieve sterilization or reinsertion to achieve IUD placement
Reoperation to achieve sterilization or reinsertion to achieve IUD placement | 12 months post-procedure
  Evaluating rates of reoperation to achieve sterilization or reinsertion to achieve IUD placement
Reoperation to achieve sterilization or reinsertion to achieve IUD placement | 24 months post-procedure
  Evaluating rates of reoperation to achieve sterilization or reinsertion to achieve IUD placement
Reoperation to achieve sterilization or reinsertion to achieve IUD placement | 36 months post-procedure
  Evaluating rates of reoperation to achieve sterilization or reinsertion to achieve IUD placement
Reoperation to achieve sterilization or reinsertion to achieve IUD placement | 48 months post-procedure
  Evaluating rates of reoperation to achieve sterilization or reinsertion to achieve IUD placement
Reoperation to achieve sterilization or reinsertion to achieve IUD placement | 60 months post-procedure
  Evaluating rates of reoperation to achieve sterilization or reinsertion to achieve IUD placement
Need for subsequent surgery to remove foreign body, remove fallopian tube(s) (salpingectomy), or uterus (hysterectomy) | 3 months post-procedure
  Need for surgical procedure after hysteroscopic or laparoscopic sterilization or IUD placement as assessed by surgery to remove foreign body, salpingectomy, or hysterectomy
Need for subsequent surgery to remove foreign body, remove fallopian tube(s) (salpingectomy), or uterus (hysterectomy) | 6 months post-procedure
  Need for surgical procedure after hysteroscopic or laparoscopic sterilization or IUD placement as assessed by surgery to remove foreign body, salpingectomy, or hysterectomy
Need for subsequent surgery to remove foreign body, remove fallopian tube(s) (salpingectomy), or uterus (hysterectomy) | 12 months post-procedure
  Need for surgical procedure after hysteroscopic or laparoscopic sterilization or IUD placement as assessed by surgery to remove foreign body, salpingectomy, or hysterectomy
Need for subsequent surgery to remove foreign body, remove fallopian tube(s) (salpingectomy), or uterus (hysterectomy) | 24 months post-procedure
  Need for surgical procedure after hysteroscopic or laparoscopic sterilization or IUD placement as assessed by surgery to remove foreign body, salpingectomy, or hysterectomy
Need for subsequent surgery to remove foreign body, remove fallopian tube(s) (salpingectomy), or uterus (hysterectomy) | 36 months post-procedure
  Need for surgical procedure after hysteroscopic or laparoscopic sterilization or IUD placement as assessed by surgery to remove foreign body, salpingectomy, or hysterectomy
Need for subsequent surgery to remove foreign body, remove fallopian tube(s) (salpingectomy), or uterus (hysterectomy) | 48 months post-procedure
  Need for surgical procedure after hysteroscopic or laparoscopic sterilization or IUD placement as assessed by surgery to remove foreign body, salpingectomy, or hysterectomy
Need for subsequent surgery to remove foreign body, remove fallopian tube(s) (salpingectomy), or uterus (hysterectomy) | 60 months post-procedure
  Need for surgical procedure after hysteroscopic or laparoscopic sterilization or IUD placement as assessed by surgery to remove foreign body, salpingectomy, or hysterectomy
Number of participants with new onset chronic pain as assessed by new prescriptions for narcotics | 3 months post-procedure
  New prescription for narcotics after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset chronic pain as assessed by new prescriptions for narcotics | 6 months post-procedure
  New prescription for narcotics after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset chronic pain as assessed by new prescriptions for narcotics | 12 months post-procedure
  New prescription for narcotics after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset chronic pain as assessed by new prescriptions for narcotics | 24 months post-procedure
  New prescription for narcotics after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset chronic pain as assessed by new prescriptions for narcotics | 36 months post-procedure
  New prescription for narcotics after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset chronic pain as assessed by new prescriptions for narcotics | 48 months post-procedure
  New prescription for narcotics after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset chronic pain as assessed by new prescriptions for narcotics | 60 months post-procedure
  New prescription for narcotics after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset depression as assessed by new prescriptions for antidepressants | 3 months post-procedure
  New prescription for anti-depressant medication after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset depression as assessed by new prescriptions for antidepressants | 6 months post-procedure
  New prescription for anti-depressant medication after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset depression as assessed by new prescriptions for antidepressants | 12 months post-procedure
  New prescription for anti-depressant medication after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset depression as assessed by new prescriptions for antidepressants | 24 months post-procedure
  New prescription for anti-depressant medication after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset depression as assessed by new prescriptions for antidepressants | 36 months post-procedure
  New prescription for anti-depressant medication after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset depression as assessed by new prescriptions for antidepressants | 48 months post-procedure
  New prescription for anti-depressant medication after hysteroscopic compared to laparoscopic sterilization and IUD placement
Number of participants with new onset depression as assessed by new prescriptions for antidepressants | 60 months post-procedure
  New prescription for anti-depressant medication after hysteroscopic compared to laparoscopic sterilization and IUD placement
Pre-procedure clinical variables associated with procedural complications | Up to 1-year pre-procedure
  Identify sociodemographic and pre-procedure clinical variables which may predict complications following hysteroscopic sterilization compared to laparoscopic sterilization and IUD placement

CONTACTS AND LOCATIONS:
Overall Officials: Aileen Gariepy, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gariepy AM, Lewis C, Zuckerman D, Tancredi DJ, Murphy E, McDonald-Mosley R, Sonalkar S, Hathaway M, Nunez-Eddy C, Schwarz EB. Comparative effectiveness of hysteroscopic and laparoscopic sterilization for women: a retrospective cohort study. Fertil Steril. 2022 Jun;117(6):1322-1331. doi: 10.1016/j.fertnstert.2022.03.001. Epub 2022 Apr 12. PMID 35428480
- [Derived] Schwarz EB, Lewis CA, Dove MS, Murphy E, Zuckerman D, Nunez-Eddy C, Tancredi DJ, McDonald-Mosley R, Sonalkar S, Hathaway M, Gariepy AM. Comparative Effectiveness and Safety of Intrauterine Contraception and Tubal Ligation. J Gen Intern Med. 2022 Dec;37(16):4168-4175. doi: 10.1007/s11606-022-07433-4. Epub 2022 Feb 23. PMID 35194746
- [Derived] Gariepy AM, Lewis C, Zuckerman D, Tancredi DJ, Murphy E, McDonald-Mosley R, Sonalkar S, Hathaway M, Nunez-Eddy C, Schwarz EB. Patient-Centered Safety Outcomes After Hysteroscopic Compared With Laparoscopic Sterilization. Obstet Gynecol. 2022 Mar 1;139(3):423-432. doi: 10.1097/AOG.0000000000004690. PMID 35115444
- See also: This work was (partially) supported through a Patient-Centered Outcomes Research Institute (PCORI) Award 1609-36359 — https://www.pcori.org/research-results/2017/real-world-effectiveness-and-safety-hysteroscopic-essure%C2%AE-compared